CLINICAL TRIAL: NCT03513653
Title: Strain for Risk Assessment and Therapeutic Strategies in Patients With Acute Heart Failure (STRATS-AHF) Registry
Acronym: STRATS-AHF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Goo-Yeong Cho, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1702/384-111
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure Acute; Heart Failure; Echocardiography
Keywords: acute heart failure; global longitudinal strain; ejection fraction; echocardiography; mortality
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute heart failure: Patients hospitalized for acute heart failure and underwent echocardiography with speckle-tracking imaging
  Interventions: Diagnostic Test: Echocardiography with speckle-tracking imaging

INTERVENTIONS:
Diagnostic Test: Echocardiography with speckle-tracking imaging — 1. Measurement of left ventricular ejection fraction and global longitudinal strain
  2. Measurement of left atrial reservoir strain (peak atrial longitudinal strain)
  3. Measurement of right ventricular global longitudinal strain

SUMMARY:
STRATS-AHF (STrain for Risk Assessment and Therapeutic Strategies in patients with Acute Heart Failure) registry enrolled 4,312 patients hospitalized for acute HF from 3 tertiary university hospitals (Seoul National University Bundang Hospital, Seoul National University Hospital, and Chungnam National University Hospital) from January 2009 through December 2016.

DETAILED DESCRIPTION:
Patients with signs or symptoms of heart failure and either lung congestion, or objective findings of left ventricular (LV) systolic dysfunction or structural heart disease, were eligible for the study. Echocardiography was performed and both LV ejection fraction (LVEF) and LV global longitudinal strain (LV-GLS), right ventricular GLS (RV-GLS) were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs or symptoms of HF and either lung congestion, or objective findings of LV systolic dysfunction or structural heart disease

Exclusion Criteria:

* Patients who presented with acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute heart failure
Sampling Method: Probability Sample
Enrollment: 4312 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | up to 5 years
  Death from any cause

SECONDARY OUTCOMES:
Hospitalization for heart failure | up to 5 years
  Any hospitalization for acute heart failure after the index hospitalization
Composite of all-cause mortality and hospitalization for heart failure | up to 5 years
  Death from any cause or any hospitalization for acute heart failure after the index hospitalization
Ischemic stroke | up to 5 years
  Ischemic stroke (an episode of neurological dysfunction caused by embolism) after the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Goo-Yeong Cho, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park JJ, Park JB, Park JH, Cho GY. Global Longitudinal Strain to Predict Mortality in Patients With Acute Heart Failure. J Am Coll Cardiol. 2018 May 8;71(18):1947-1957. doi: 10.1016/j.jacc.2018.02.064. PMID 29724346
- [Background] Park JH, Park JJ, Park JB, Cho GY. Prognostic Value of Biventricular Strain in Risk Stratifying in Patients With Acute Heart Failure. J Am Heart Assoc. 2018 Oct 2;7(19):e009331. doi: 10.1161/JAHA.118.009331. PMID 30371332
- [Background] Hwang IC, Cho GY, Choi HM, Yoon YE, Park JJ, Park JB, Park JH, Lee SP, Kim HK, Kim YJ, Sohn DW. Derivation and validation of a mortality risk prediction model using global longitudinal strain in patients with acute heart failure. Eur Heart J Cardiovasc Imaging. 2020 Dec 1;21(12):1412-1420. doi: 10.1093/ehjci/jez300. PMID 31819981
- [Background] Park JJ, Choi HM, Hwang IC, Park JB, Park JH, Cho GY. Myocardial Strain for Identification of beta-Blocker Responders in Heart Failure with Preserved Ejection Fraction. J Am Soc Echocardiogr. 2019 Nov;32(11):1462-1469.e8. doi: 10.1016/j.echo.2019.06.017. Epub 2019 Sep 17. PMID 31540679
- [Background] Park JH, Hwang IC, Park JJ, Park JB, Cho GY. Prognostic power of left atrial strain in patients with acute heart failure. Eur Heart J Cardiovasc Imaging. 2021 Jan 22;22(2):210-219. doi: 10.1093/ehjci/jeaa013. PMID 32031588
- [Background] Park CS, Park JB, Park JJ, Park JH, Cho GY. Impact of sex and myocardial function on association of obesity with mortality in Asian patients with acute heart failure: a retrospective analysis from the STRATS-AHF registry. BMJ Open. 2020 Feb 10;10(2):e031608. doi: 10.1136/bmjopen-2019-031608. PMID 32047009
- [Background] Park JJ, Mebazaa A, Hwang IC, Park JB, Park JH, Cho GY. Phenotyping Heart Failure According to the Longitudinal Ejection Fraction Change: Myocardial Strain, Predictors, and Outcomes. J Am Heart Assoc. 2020 Jun 16;9(12):e015009. doi: 10.1161/JAHA.119.015009. Epub 2020 Jun 10. PMID 32519555
- [Background] Park JJ, Park JH, Hwang IC, Park JB, Cho GY, Marwick TH. Left Atrial Strain as a Predictor of New-Onset Atrial Fibrillation in Patients With Heart Failure. JACC Cardiovasc Imaging. 2020 Oct;13(10):2071-2081. doi: 10.1016/j.jcmg.2020.04.031. Epub 2020 Jul 15. PMID 32682715
- [Derived] Park JH, Kim M, Park JJ, Park JB, Cho GY. Prognostic Role of RVGLS/PASP Ratio, a New Echocardiographic Parameter of the Right Ventricle-Pulmonary Artery Coupling, in Patients With Acute Heart Failure. Int J Heart Fail. 2024 Oct 28;6(4):165-173. doi: 10.36628/ijhf.2024.0048. eCollection 2024 Oct. PMID 39513018
- [Derived] Park CS, Park JJ, Hwang IC, Park JB, Park JH, Cho GY. Myocardial strain to identify benefit from beta-blockers in patients with heart failure with reduced ejection fraction. ESC Heart Fail. 2022 Apr;9(2):1248-1257. doi: 10.1002/ehf2.13800. Epub 2022 Jan 9. PMID 35001562
- [Derived] Park CS, Hwang IC, Park JJ, Park JH, Park JB, Cho GY. Determinants of the survival benefit associated with statins in patients with acute heart failure. ESC Heart Fail. 2021 Dec;8(6):5424-5435. doi: 10.1002/ehf2.13637. Epub 2021 Oct 5. PMID 34612019